CLINICAL TRIAL: NCT00183937
Title: A Phase II Study of Bortezomib (Velcade®, PS-341) and Docetaxel for Patients With Hormone Refractory Prostate Cancer
Brief Title: Study of Bortezomib and Docetaxel for Patients With Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4P-04-3
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Bortezomib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib and Docetaxel (Experimental): Bortezomib 1.6 mg/m2 Docetaxel 75 mg/m2
  Interventions: Drug: PS 341; Drug: Docetaxel

INTERVENTIONS:
Drug: PS 341 — PS 341 1.6 mg/m2 IV (in the vein) on days 1 and 8 of each 21 day cycle up to 12 cycles.
  Other Names: Bortezomib; Velcade
Drug: Docetaxel — Docetaxel 75mg/m2 IV (in the vein) on day 1 of each 21 day cycle up to 12 cycles.

SUMMARY:
This study is for patients who have been treated with surgical removal of the testes or hormone therapy (Lupron or Zoladex) and whose prostate cancer has worsened despite this treatment.

PS 341 is a type of drug known as a "proteasome inhibitor." By inhibiting the "proteasome" in cancer cells, PS-341 alters the way those cells divide). We hope to learn whether this combination chemotherapy decreases cancer symptoms and tests (prostate specific antigen, also called PSA), and to determine how frequently serious side effects might occur with this treatment for this stage of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have had a histological or cytological diagnosis of adenocarcinoma of prostate and currently must have metastatic disease (stage TxNxM1) that is unresponsive or refractory to hormone therapy. Patients must have metastatic prostate cancer deemed to be hormone refractory by one or more of the following (despite androgen ablation and anti-androgen withdrawal where applicable):
* Progression of measurable disease assessed within 28 days prior to registration. OR
* Progression of non-measurable (i.e. bone scan or PET scan) disease assessed within 42 days prior to registration. AND
* Rising PSA - defined as at least 2 consecutive rises in PSA documented over a reference value (measure 1). The first rising PSA (measure 2) should be taken at least 7 days after the reference value. A third confirmatory PSA measure is required (2nd beyond the reference level) to be greater then the second measure and it must be obtained at least 7 days after the 2nd measure. Patient must have a PSA concentration of at least 5 ng/ml in addition to increasing PSA to be eligible Note: The PSA result (done within 28 days prior to registration) need not be elevated for inclusion provided other criteria for progression are met and the serum PSA is at least 2 ng/ml.
* Must have received prior hormonal therapy and have a castrate level of testosterone (less than 100ng/ml within 90 days of entry to the study). Patients treated with orchiectomy are eligible. If patients have been treated with non-steroidal anti-androgens, the patients must have ceased taking flutamide or nilutamide at least 28 days prior to enrollment and at least 42 days prior to enrollment for biclutamide. Either method of castration can have been supplemented with nonsteroidal antiandrogen (e.g. flutamide, biclutamide, nilutamide). Patients may have been treated with "second-line" hormonal therapy such as ketoconazole, aminoglutethimide and/or estrogen therapies but these must have ceased at least 7 days prior to commencement of study therapy.
* May have received at most one prior chemotherapy for hormone refractory prostate cancer provided they have not received docetaxel or Bortezomib for that indication or otherwise within 2 years of trial entry.
* Prior radiation therapy is allowed but it must have been to less than 25% of total body bone marrow. This includes prior use of samarium, but patients can not have received strontium. (>10 days must have elapsed since completion of RT with recovery from side effects. Soft tissue disease irradiated in the prior 2 months is not and may not be designated as measurable
* Creatinine less than or equal to 1.5x the institutional upper limit of normal (within 28 days prior to registration)
* Hepatic function Total Bilirubin less than or equal to ULN AST and ALT and Alkaline Phosphatase must be within the range allowing for eligibility.

In determining eligibility the more abnormal of the two values (AST or ALT) should be used.

* Adequate bone marrow function. Complete blood count with differential must be done within 14 days prior to registration Absolute neutrophil count greater than or equal to 1,500/mm3 Hemoglobin greater than or equal to 8.0 g/dl Platelet count greater than or equal to 100,000/mm3
* ECOG performance status 0-3. (For patients with PS of 3, cause must be due to pain secondary to bone metastases to be eligible)
* Patients should (for good medical practice) have stabilization of their analgesic medications for at least one week prior to receiving study medication
* No other chemotherapy, biological response modifiers, RT, radioisotope therapy (e.g. samarium or strontium), corticosteroid, or concomitant hormonal therapy may be given during protocol treatment.
* Bisphosphonate therapy is permitted provided it commences prior to study entry and is maintained at recommended dosing intervals.
* Completed baseline McGill Pain Questionnaire and Pain Medication Log prior to registration. The nurse or CRA must complete MPQ and PML cover sheet for baseline assessment prior to registration. If unable to complete questionnaires in English or Spanish, patient can be registered without contributing to QOL study).
* Men of childbearing potential must be willing to consent to using effective contraception while on treatment and for a reasonable period (90 days) thereafter.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* Myocardial infarction or angina pectoris within one year of registration
* History of brain metastases, treated or untreated. (Patients with neurological symptoms must have CT or MRI brain negative for metastatic disease within 56 days prior to registration). Patients who have recovered from spinal cord compression and are clinical stable may enter the study provided they fulfill other criteria.
* Not recovered from major infections and/or surgical procedures, or has significant active concurrent other medical illness precluding protocol therapy or survival.
* Known or anticipated severe hypersensitivity reaction to bortezomib, boron, mannitol, docetaxel or polysorbate 80.
* Other prior malignancy (except patients who have had another stage I or II malignancy currently in complete remission or other cancer with no evidence of disease for greater than 5 years from accrual to the current trial. Patients with basal or squamous cell carcinoma of the skin that have been treated with curative intent can be accrued to this trial 30 days after treatment. Solar keratoses treated topically do not preclude entry).
* Patient has greater than or equal to Grade 2 peripheral neuropathy within 14 days before enrollment.
* Prior therapy with docetaxel or paclitaxel
* Prior treatment with more than one prior chemotherapy for hormone refractory prostate cancer.
* Ongoing therapy with drugs known to inhibit P4503A4 drug metabolism including:

Macrolide antibiotics: erythromycin, troleandomycin, azithromycin Imidazole antifungal agents: ketoconazole, itraconazole, fluconazole HIV protease inhibitors Immunosuppressive agents: cyclosporin, FK-506

* Ongoing therapy with drugs known to induce P4503A4 drug metabolism including: Phenobarbital, phenytoin, carbamazepine, griseofuvin and rifampin.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-04-30 (Actual); Primary Completion 2010-10-23 (Actual); Study Completion 2012-06-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with improved serum PSA response rate | Every end of each cycle (21 days) up to 12 cycles
  Participants should be reevaluated for PSA response every 21 days. A confirmatory PSA level should be obtained 3-4 weeks following initial documentation of a PSA response.

SECONDARY OUTCOMES:
Pain response rate | At baseline, then weekly for 4 weeks up to 36 weeks
  Participants will be considered evaluable for a pain response if the baseline analgesic use was determined, and at least 4 weekly assessments of PPI and analgesic score are available from any 8-week period from the period after the initiation of therapy until discontinuation of study medication.

CONTACTS AND LOCATIONS:
Overall Officials: David Quinn, MD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States